CLINICAL TRIAL: NCT03308994
Title: Impact of the Arrival on the French Market of New First Line Oral Treatments on the Delay Between MS Onset and First Disease Modifying Treatment (DMTs) Administration
Acronym: PREMISEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 16-913
Record Dates: First submitted 2017-08-18; First posted 2017-10-13 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: C10.114.375.500
Keywords: Multiple sclerosis; Epidemiology; Oral disease modifying treatments; Therapeutical delays; Socio-Economic Status
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral first line disease modifying treatments
  Interventions: Other: Delay between MS onset and introduction of first line DMT; Other: EDI
- Injectable first line disease modifying treatments
  Interventions: Other: Delay between MS onset and introduction of first line DMT; Other: EDI

INTERVENTIONS:
Other: Delay between MS onset and introduction of first line DMT — Delay between MS onset and introduction of first line DMT : time between date of MS onset ( the first demyelinating neurological events clinically defined) and date of the introduction of the first-line oral DMT (Interferons, Glatiramer Acetate, Dimethyl Fumarate and Teriflunomide)
Other: EDI — For all cases of multiple sclerosis residence's places of each patient were geolocalized with a Geographic Information System (ARCGIS 10.2) and assigned to an IRIS, IRIS (Ilots Regroupés pour l'Information Statistique) is the smallest French geographic unit for which census data are available and EDI score was calculated for each IRIS. In order to attribute a social deprivation score to the IRIS, we used the French EDI (European Deprivation Index). EDI stands as a continuous variable but EDI will be used as a categorical variable in order to increase the comparability with others studies, so EDI is distributed into quintiles calculated at the French level.

SUMMARY:
The study design matches with a multicenter observational ambispective study. A first pilot study will be undertaken in Caen center and is expected to be extended to Rouen and Lille center. So patients from Normandy and North-West areas will be included.

In order to include patients in this observational study historical data about first line injectable treatments (interferons and glatiramer acetate) are used. As well as the data on patients treated with oral first line therapies (teriflunomide and dimethyl fumarate) began to be collected ahead of the study start (Retrospective phase). During the course of the study, new patients under teriflunomide or dimethyl fumarate will be included (Prospective phase).

DETAILED DESCRIPTION:
Multiple sclerosis is known to be the first non traumatic cause of disability in young people. Multiple sclerosis is described as a chronic inflammatory immune-mediated disease of the central nervous system.

Only a few disease modifying treatments where available before 1994, but in two decades, the therapeutic armamentarium was reinforced by many more and more effective drugs for RRMS .They tend to extend time to conversion towards a defined MS after the first relapse and between relapses and have a notable action on the decreasing clinical and radiological disease activity.

First line of disease modifying treatments (DMTs), IFN β-1a and glatiramer acetate are known to have a favorable benefit-to-risk profile in RRMS, they reduce relapse rate and MRI activity of the disease, but their efficacy remains limited. They do not stop the disease progression but only slow down it for a while. Otherwise four drugs cyclophosphamide, mitoxantrone, natalizumab and fingolimod were used as second-line therapy or as first-line for rapidly evolving RRMS. Whereas second line DMTs cyclophosphamide and mitoxantrone were merely an alternative to pharmacological run away, natalizumab and fingolimod proved to be two effective drugs of second line DMTs. Natalizumab impressively inhibits inflammatory process of MS, with >65% reduction in relapses during 2 years of treat¬ment, and >90% suppression of new inflammatory MRI lesions and fingolimod suppresses MS disease activity with 55-60% of lower relapses rates and a remarkable decrease of visible MRI activity . In 2014 alemtuzumab received FDA approval and joined the other second line treatment but it is still not commercialized in France. Recently years two new first line treatments teriflunomide and dimethyl fumarate have made their entry on the market. The main advantage of these both treatments is their mode of administration. Whereas the two first line treatments are under injectable form, teriflunomide and dimethyl fumarate can be administered per os, and so facilitate the therapy compliance for newly-diagnosed RRMS patients. In TEMSO, a phase III multicentric double-blinded study with teriflunomide 14 mg once a day versus placebo, teriflunomide shows both efficacy in reducing from 31,5% relapse rate in 2 years and a significant 80.4% of reduction of MRI activity for T1 enhanced lesions by gadolinium. Risk of disability progression is also significantly reduced of 29.8%, as compared with placebo. Efficacy and safety phase 3 trial study DEFINE assessed efficacy of BG-12 (dimethyl fumarate) 240 mg given orally either twice daily significantly reduced the risk of relapse by 49% or compared with placebo at 2 years. On ARR, there were relative reductions of 53% .The probability of confirmed 12-week disability progression was reduced by 38%. In an MRI sub-study the mean number of new or newly enlarging T2 lesions was reduced by 85% . A clear efficacy on disease activity is shown when comparing respectively dimethylfumarate and teriflunomide with placebo.

However the efficacy on clinical symptoms and disease activity isn't significantly better than that of the first line's treatments of references. Compare to glatiramer acetate, dimethyl fumarate shows no significant greater clinical effect on the disease . No significant annual relapses rate difference was shown either between teriflunomide and interferon ß-1a . The most interesting progress of these two molecules lies in their easier mode of administration and the inherent change of medical practices.

Diagnosis and therapeutic delays have already proved to be some remarkable health indicators in numerous chronic or serious diseases. In cancers, "diagnostic delays" and "therapeutics delays" are demonstrated to have an negative impact survival and mortality . Various delays may occur at different stages of health care. On the one hand diagnosis delays are a complex association of "patients delay" (from onset of symptoms to their first presentation), depending on patients factors as behavior or social background, "referral delay" (from general practician's medical consultation to a specialist one), and finally "delay to lead a diagnosis" (time required to undergo specialized medical examinations). On the other hand therapeutics delays (from diagnosis to start of the treatment) are more associated with health system process (15,16).

Evolution of diagnosis criteria and especially last revision of McDonald 2010 criteria, that show high sensibility and specificity, obviously influence healthcare delays by allowing early diagnosis and indirectly early treatment initiation. .

Treatment delays are also shorten by the evidence of a favorable impact of early treatment initiation for patients with RRMS . Early DMT initiation seems to be beneficial for MS patients. Early treatment with INF-1b reduced the risk of clinically determined Multiple Sclerosis (CDMS) by 37% compared with delayed treatment after a 5 year follow-up . Early treatment with glatiramer acetate is efficacious in delaying conversion to CDMS in patients presenting with clinically isolated symptoms (CIS) and brain lesions detected by MRI. Time for 25% of patients to convert to CDMS was prolonged from 336 days for Placebo to 722 days for glatiramer acetate. Similar data have been found with early treatment with glatiramer acetate 40 mg injected 3 times a week: reductions in annual relapses rate, lesion activity, and evolution of active lesions to chronic black holes over 3 years. For new oral treatments, same significant results highlight the benefit of an early teriflunomide initiation. In an extension of TOWER study in patients receiving teriflunomide 14 mg for up to 5.5 years, comparisons of early versus s delayed treatment initiation was made. An estimated 26.7% of patients in the early treatment group experienced disability progression confirmed for ≥12 weeks versus an estimated 30.2% in the delayed treatment group. Moreover a relative reduction of 29.9% of annual relapses rate was significantly proved between early treatment group and the delayed treatment group. And time of first relapse is significantly longer in the early treatment group than in the delayed one.

Social determinants in public health issues have interested worldwide many researchers, and international comparisons show that social inequalities in health are particularly pronounced in France despite a global good quality health system.

Previous studies in the US have found that depending on insurance status and social position (education, employment status ) there were a difference in accessing specialty MS care . Patients followed by MS multidisciplinary network benefit of a better global care, they are more likely to undergo diagnosis tests and be prescribed DMT's. As patients socially deprived have a limited access to MS multidisciplinary network, they benefit of a lower global health care quality.

In survey studies lead in 50 states of the United Sates significant differences appears between urban/rural on residency in accessing specialty MS care providers. MS patients who live in more remote rural areas received MS focused areas at the same place than their routine health care, whereas their urban counterparts have an easier access to MS clinics or MS health centers. Most of geographically isolated patients haven't recourse to MS related cares because of greater travel times to receive MS care from specialist (27). There are differences in the use of physician services patients according to urban or rural on residency. In more remote rural areas one on three patients does not consult a neurologist or MS specialist as much as they would like. Patients who lives in rural areas do not received the same appropriate MS focused cares than their urban counterparts . Distances and travel times to access MS related cares may also act as a loss of chances for patients.

In the last two decades, there was a progressive evolution of therapies and every new drugs type arrival on the market being synonymous of medical practices evolutions and patients healthcare. First line oral DMT(s) obviously represent an improvement in ease of treatments' administration. So an impact of the recent treatments teriflunomide and dimethyl fumarate arrival in reducing therapeutic healthcare delays can be hypothesized.

Addition to complete this study, a second hypothesis can be formulated. Social inequalities and geographic disparities strongly have an impact on patients medical and treatment initiation, so improving drug delivery will probably moderate this impact.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered in EDMUS database.
* Patients with an initial and definite diagnosis of Relapsing-Remitting Multiple Sclerosis.
* An established diagnosis from January 1st 1995 to the end of the study.

Exclusion Criteria:

* Patients not registered in EDMUS database.
* Patient with a diagnosis of Primary Progressive Multiple Sclerosis
* Patients with a diagnosis established before January 1st 1995

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: RRMS patients treated with oral or injectable first line DMT.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Date of MS onset | From date of the first neurological event to the end of the study in december 2018, as only date after 1982 were retained the time frame is up to 36 years.
  Date of the first neurological event. Only the date of MS onset after 1982 were retained.
Date of introduction of first line DMT | From date of the primo-prescription of a first injectable or oral first line DMT to the end of the study in december 2018. The time frame is up to 23 years.
  Date of the primo-prescription of a first injectable or oral first line DMT.
Residence location | To calculate EDI scores, addresses' of patients were required and were collected since EDMUS base was operational in 2004 until the end of the study. The time frame is up to 14 years.
  For all cases of multiple sclerosis residence's places of each patient were geo-localized with a Geographic Information System (ARCGIS 10.2) and assigned to an IRIS, IRIS (Ilots Regroupés pour l'Information Statistique) is the smallest French geographic unit for which census data are available and EDI score was calculated for each IRIS. In order to attribute a social deprivation score to the IRIS, we used the French EDI (European Deprivation Index). EDI stands as a continuous variable but EDI will be used as a categorical variable in order to increase the comparability with others studies, so EDI is distributed into quintiles calculated at the French level. EDI stands as a continuous variable but EDI will be used as a categorical variable in order to increase the comparability with others studies, so EDI is distributed into quintiles calculated at the French level.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Groupement des Hôpitaux de l'Institut Catholique de Lille (HICL), Lille, Hauts-de-France
  - University Hospital of Lille, Lille, Hauts-de-France
  - University Hospital Center of Caen, Caen, Normandy
  - University Hospital of Rouen, Rouen, Normandy

IPD SHARING:
Plan to Share IPD: No